CLINICAL TRIAL: NCT00362310
Title: A Phase II Trial With the HIV Protease Inhibitor Indinavir for the Treatment of Classical Kaposi's Sarcoma
Brief Title: Treatment of Classical Non-HIV-Related Kaposi's Sarcoma With the Antiviral Drug Indinavir
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Istituto Superiore di Sanità (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CKS/IND/02
Record Dates: First submitted 2006-08-09; First posted 2006-08-10 (Estimated); Last update posted 2008-04-14 (Estimated); Status verified 2008-04

CONDITIONS: Classical Kaposi's Sarcoma
Keywords: classical kaposi's sarcoma; treatment; HIV protease inhibitor indinavir
MeSH Terms: interventions — Indinavir

INTERVENTIONS:
Drug: indinavir

SUMMARY:
Recent studies have described a reduced incidence or the regression of Kaposi's sarcoma (KS) in HIV-infected patients treated with the highly active anti-retroviral therapy (HAART) that contains at least one inhibitor of the HIV protease (HIV-PI) such as Indinavir. Experimental studies have shown that part of the anti-KS actions of HIV-PI are not related to their antiretroviral actions, but, at least in part, to their capability of blocking angiogenesis and tumor growth.

This study will be conducted on HIV-negative (classical) KS patients to prove that Indinavir has anti-angiogenic and anti-KS effects in humans independently of its antiretroviral activity.

DETAILED DESCRIPTION:
Kaposi's sarcoma (KS) is a rare vascular tumor affecting elderly individuals from Mediterranean countries (CKS), post transplant patients and, with increased incidence and aggressiveness, HIV-infected individuals (AIDS-KS). No definitive cure has been established for KS and all conventional therapies result in low response rate, high toxicity and tumor relapse.

Antiretroviral therapies including a HIV protease inhibitor (HIV-PI) have reduced AIDS-KS incidence and induce KS regression in treated patients. This cannot be explained solely with drug-mediated HIV suppression and immune reconstitution. We have shown that HIV-PI such as Indinavir or Saquinavir block KS-like lesions in mice by inhibiting angiogenesis and tumor cell invasion through a blockade of matrix metalloprotease 2 (MMP2) proteolytic activation.

Based on these data, a proof-of-concept clinical study on HIV-negative (classic) KS (C-KS) patients was planned to prove that Indinavir has anti-angiogenic and anti-KS effects in humans independently of its antiretroviral activity.

Recent concepts in the evaluation of non cytotoxic anti-cancer drugs such as anti-angiogenic agents suggest novel criteria for the design of clinical studies due to the specific mechanism of action of these drugs. In particular, the use of the conventional evaluation criteria based on cytotoxic actions may mislead the interpretation of the therapeutic efficacy of non cytotoxic agents. The study was therefore designed to compare the clinical response to Indinavir in early-stage vs. late-stage KS and by relating it to key biological endpoints and plasmatic drug concentrations. This was also motivated by the rareness of C-KS and by ethical reasons which prevented the inclusion of a control group.

Patients will be treated per os with 800 mg x 2/daily of Indinavir for 12 months. Follow-up will be one year.

Primary objectives:

Evaluation of the tumor response rate (complete response, partial response, improved disease and stable disease) to indinavir in the treatment of mild or severe classical KS patients; Evaluation of the duration of response in indinavir-treated patients.

Secondary objectives:

Evaluation of Indinavir safety in classical KS population; Determination of the pharmacokinetic profile of Indinavir; Evaluation of key Kaposi's sarcoma biological endpoints including markers of angiogenesis and tumor invasion, Th1 and Th2 polarization of the immune response, immunoactivation, and immune responses to HHV8, herpesviruses and common pathogens.

ELIGIBILITY:
Inclusion Criteria:

* Have a documented diagnosis of classical KS
* Be HIV-negative
* Be 18 years old and over
* Have one or more of the following: a minimum of 3 measurable progressive lesions; all stages of complicated KS, i.e. showing functional impotency of the affected limbs, lymphedema, lymphorrea or pain; visceral disease; lack of response to conventional therapy (radiotherapy, chemotherapy); contraindication to conventional therapies-

Exclusion Criteria:

* Presence of life-threatening lesions or other concomitant illness, neoplasia or any other clinical condition threatening the health of the patient or his compliance to the treatment
* Inability to provide informed consent
* Concomitant treatment (within 30 days of initiating study treatment) with systemic immunomodulatory agents (e.g., glucocorticoids as immunosuppressive agents, interferons) or chemotherapy
* Pregnancy
* Impaired clinical conditions (Karnofsky's index <60
* Diabetes, history of nephrolithiasis or monolateral nephropathy
* Difficulty swallowing capsules/tablets
* Any clinically significant laboratory findings obtained during screening, including:

  * Alkaline phosphatase (AP) >2 fold upper limit of normal (ULN)
  * Aspartate aminotransferase (AST)
  * Alkaline aminotransferase (ALT)
  * Gamma-glutamyl transferase (gamma-GT) or total bilirubin >3 fold the ULN
  * Serum creatinine >1.2 mg/d for women and >1.4 mg/dL for men or creatinine clearance > 100 +/- 25
  * Pancreatic amylase >1.5 folds ULN
  * Hemoglobin <10.0 g/dL for males, <9.0 g/dL for females
  * Platelet count <75.000/cubic millimeter (mm3)
  * Neutrophil count <850/mm3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28
Dates: Start 2003-06; Study Completion 2007-07

PRIMARY OUTCOMES:
Assessment of clinical response every 3 months during treatment and every 6 months during follow-up based on the recommendations of ACTG.

SECONDARY OUTCOMES:
Monthly evaluation of toxicity and of biological endpoints every 3 months and their correlation with drug plasma levels

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Ensoli, MD, PhD, Study Chair — National AIDS Center, Istituto Superiore di Sanità, Rome, Italy
Locations (9):
- Italy (9):
  - Centro di Riferimento Oncologico (CRO),, Aviano
  - Department of Internal Medicine, University of Cagliari, Cagliari
  - Dermatologic Clinic, Ospedale S. Anna, Ferrara
  - Ospedale Maggiore, Mangiagalli e Regina Elena, IRCCS,, Milan
  - Ospedale Civico Benfratelli, Palermo
  - Department of Dermatological/Venereal Diseases and Plastic Surgery, University "La Sapienza", Rome
  - Istituto Dermatologico S. Gallicano-IRCCS, Rome
  - Istituto Dermopatico dell'Immacolata-IRCCS (IDI), Rome
  - Dermatology Clinic, University of Sassari, Sassari

REFERENCES:
- [Background] Monini P, Sgadari C, Toschi E, Barillari G, Ensoli B. Antitumour effects of antiretroviral therapy. Nat Rev Cancer. 2004 Nov;4(11):861-75. doi: 10.1038/nrc1479. PMID 15516959
- [Background] Sgadari C, Barillari G, Toschi E, Carlei D, Bacigalupo I, Baccarini S, Palladino C, Leone P, Bugarini R, Malavasi L, Cafaro A, Falchi M, Valdembri D, Rezza G, Bussolino F, Monini P, Ensoli B. HIV protease inhibitors are potent anti-angiogenic molecules and promote regression of Kaposi sarcoma. Nat Med. 2002 Mar;8(3):225-32. doi: 10.1038/nm0302-225. PMID 11875492